CLINICAL TRIAL: NCT01074229
Title: The Effect of Pre-operative Transversus Abdominis Plane (TAP) Block in the Quality of Recovery of Patients Undergoing Laparoscopic Hysterectomy: a Prospective, Randomized, Blinded Study
Brief Title: Transversus Abdominis Plane (TAP) Block Laparoscopic Hysterectomy
Acronym: TAP HYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00023440
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Postoperative Pain
Keywords: Pain; Post Operative; Opioids; Laparoscopic; Surgery; Hysterectomy
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Pharmaceutical Preparations; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): sterile normal saline as placebo
  Interventions: Drug: Placebo
- Drug .5% Ropivacaine (Active Comparator): Instillation of 20 cc of 0.5% ropivacaine
  Interventions: Drug: Drug .5% Ropivacaine
- 20 cc of 0.25% ropivacaine (Active Comparator): Instillation of 20 cc of 0.25% ropivacaine
  Interventions: Drug: 20 cc of 0.25% ropivacaine

INTERVENTIONS:
Drug: Placebo — placebo injection
  Other Names: Sterile normal saline
  Arms: Placebo
Drug: Drug .5% Ropivacaine — .5% ropivacaine 20 mls on each side of abdomen
  Other Names: .5% Ropivacaine
  Arms: Drug .5% Ropivacaine
Drug: 20 cc of 0.25% ropivacaine — Will receive a bilateral TAP block using 20 cc of 0.25% ropivacaine
  Other Names: .25% ropivacaine
  Arms: 20 cc of 0.25% ropivacaine

SUMMARY:
The transversus abdominis plane (TAP) block involves the sensory nerve supply of the anterior -lateral abdominal wall where the T7-12 intercostal nerves, ilioinguinal, iliohypogastric and the lateral cutaneous branches of the dorsal rami of L1-3 are blocked with an injection of local anesthetic between the internal oblique abdominal muscle (IOAM) and the transverse abdominal muscle(TAM)This technique allows sensory blockade of the anterolateral abdominal wall via local anesthetic deposition superficial to the transversus abdominis muscle. It was first described by McDonnell et al. as a landmark technique to provide analgesia for lower abdominal surgery.

Hebbart et al. subsequently described an ultrasound guided technique for the TAP block which they named posterior TAP block. The ultrasound allows identification of the external oblique abdominal muscles (EOAM),IOAM and TAM. Previous studies about ultrasound -guided regional anesthetic techniques suggest improved block quality and safety, which is primarily due to direct visualization of the relevant anatomy, the tip of the needle, and the spread of the local anesthetics.

Clinical trials of the single shot posterior TAP block have shown a significant reduction in morphine consumption during the first 24-36 hours after surgery. More recently, El-dawlatly et al. demonstrated that ultrasound guided TAP block in patients undergoing laparoscopic cholecystectomy reduced perioperative opioid consumption by more than 50%.

This is the first study to evaluate the effect of TAP block in the quality of recovery in patients undergoing laparoscopic hysterectomy and may help the pathway to make this an outpatient procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-64 years
* Surgery: Laparoscopic Hysterectomy surgery
* ASA status: I and II
* Fluent in English

Exclusion Criteria:

* History of allergy to local anesthetics
* History of chronic opioid use
* Pregnant patients
* BMI greater than 30

Drop-out criteria:

* Patient or surgeon request
* Complications related to the procedure

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio DeOliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Jacobson GF, Shaber RE, Armstrong MA, Hung YY. Hysterectomy rates for benign indications. Obstet Gynecol. 2006 Jun;107(6):1278-83. doi: 10.1097/01.AOG.0000210640.86628.ff. PMID 16738152
- [Background] Babalola EO, Bharucha AE, Schleck CD, Gebhart JB, Zinsmeister AR, Melton LJ 3rd. Decreasing utilization of hysterectomy: a population-based study in Olmsted County, Minnesota, 1965-2002. Am J Obstet Gynecol. 2007 Mar;196(3):214.e1-7. doi: 10.1016/j.ajog.2006.10.390. PMID 17346525
- [Background] Lenz H, Sandvik L, Qvigstad E, Bjerkelund CE, Raeder J. A comparison of intravenous oxycodone and intravenous morphine in patient-controlled postoperative analgesia after laparoscopic hysterectomy. Anesth Analg. 2009 Oct;109(4):1279-83. doi: 10.1213/ane.0b013e3181b0f0bb. PMID 19762758
- [Background] Thiel JA, Kamencic H. Assessment of costs associated with outpatient total laparoscopic hysterectom. J Obstet Gynaecol Can. 2006 Sep;28(9):794-798. doi: 10.1016/S1701-2163(16)32258-7. PMID 17022920
- [Background] Lovatsis D, Jose JB, Tufman A, Drutz HP, Murphy K. Assessment of patient satisfaction with postoperative pain management after ambulatory gynaecologic laparoscopy. J Obstet Gynaecol Can. 2007 Aug;29(8):664-7. doi: 10.1016/s1701-2163(16)32552-x. PMID 17714620
- [Background] Wills VL, Hunt DR. Pain after laparoscopic cholecystectomy. Br J Surg. 2000 Mar;87(3):273-84. doi: 10.1046/j.1365-2168.2000.01374.x. PMID 10718794
- [Background] Goldstein A, Grimault P, Henique A, Keller M, Fortin A, Darai E. Preventing postoperative pain by local anesthetic instillation after laparoscopic gynecologic surgery: a placebo-controlled comparison of bupivacaine and ropivacaine. Anesth Analg. 2000 Aug;91(2):403-7. doi: 10.1097/00000539-200008000-00032. PMID 10910857
- [Background] Shaw IC, Stevens J, Krishnamurthy S. The influence of intraperitoneal bupivacaine on pain following major laparoscopic gynaecological procedures. Anaesthesia. 2001 Nov;56(11):1041-4. doi: 10.1046/j.1365-2044.2001.02215.x. PMID 11703235
- [Background] Moiniche S, Mikkelsen S, Wetterslev J, Dahl JB. A qualitative systematic review of incisional local anaesthesia for postoperative pain relief after abdominal operations. Br J Anaesth. 1998 Sep;81(3):377-83. doi: 10.1093/bja/81.3.377. PMID 9861124
- [Background] Keita H, Benifla JL, Le Bouar V, Porcher R, Wachowska B, Bedairia K, Mantz J, Desmonts JM. Prophylactic ip injection of bupivacaine and/or morphine does not improve postoperative analgesia after laparoscopic gynecologic surgery. Can J Anaesth. 2003 Apr;50(4):362-7. doi: 10.1007/BF03021033. PMID 12670813
- [Derived] De Oliveira GS Jr, Milad MP, Fitzgerald P, Rahmani R, McCarthy RJ. Transversus abdominis plane infiltration and quality of recovery after laparoscopic hysterectomy: a randomized controlled trial. Obstet Gynecol. 2011 Dec;118(6):1230-1237. doi: 10.1097/AOG.0b013e318236f67f. PMID 22105251

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Group B (control group) will receive sterile normal saline.
- 20 cc of 0.5% Ropivacaine: Group A (study group) 20 cc of 0.5% ropivacaine
- 20 cc of 0.25% Ropivacaine: Active Comparator 2. 20 cc of 0.25% ropivacaine
Period: Overall Study
Arm/Group | Placebo | 20 cc of 0.5% Ropivacaine | 20 cc of 0.25% Ropivacaine
Started | 25 | 25 | 25
Completed | 23 | 22 | 21
Not Completed | 2 | 3 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Change to open surgical procedure | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Study Drug: Group A (study group) 20 cc of 0.5% ropivacaine
- Total: Total of all reporting groups
Arm/Group | Placebo | Study Drug | 20 cc of 0.25% Ropivacaine | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (9.6) | 45.4 (4.5) | 46.76 (6.4) | 46.55 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 25 | 75
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: QoR40 on the Day After Surgery
Description: QoR40 on the day after surgery. Quality of recovery is based on a score of 40-200. 40 being a poor recovery and 200 being a good recovery score.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- 20 cc of 0.5% Ropivacaine: STUDY DRUG Group A (study group) 20 cc of 0.5% ropivacaine
Arm/Group | PLACEBO | 20 cc of 0.5% Ropivacaine | 20 cc of 0.25% Ropivacaine
Number analyzed (Participants) | 23 | 22 | 21
units on a scale | 152 (22.8) [136 to 167] | 180 (12.16) [169 to 190] | 180 (15.3) [161 to 184]
Statistical Analysis 1: Comparison: PLACEBO vs 20 cc of 0.5% Ropivacaine vs 20 cc of 0.25% Ropivacaine; Test type: Superiority or Other; p = .05, Kruskal-Wallis; Using Dunns test with Bonferroni conrrection for individual comparisons
Statistical Analysis 2: Comparison: PLACEBO vs 20 cc of 0.5% Ropivacaine; Test type: Superiority or Other; p = .05, Dunns test; Bonferonni correction; Median Difference (Final Values) = 28, 95% CI 2-sided [9 to 37]
Statistical Analysis 3: Comparison: PLACEBO vs 20 cc of 0.25% Ropivacaine; Test type: Superiority or Other; p = .05, Dunns Test; Bonferroni correction; Mean Difference (Net) = 28, 95% CI 2-sided [14 to 42]

2. Secondary Outcome: 24 Total Morphine Consumption
Description: Total 24 total morphine consumption post operative.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: miligrams of morphine
Arm/Group | Placebo | 20 cc of 0.5% Ropivacaine | 20 cc of 0.25% Ropivacaine
Number analyzed (Participants) | 23 | 22 | 21
miligrams of morphine | 22.75 (10.75) | 12.5 (9.84) | 17.5 (13.07)
Statistical Analysis 1: Comparison: Placebo vs 20 cc of 0.5% Ropivacaine vs 20 cc of 0.25% Ropivacaine; Test type: Superiority or Other; p = .05, Kruskal-Wallis; With Dunns test and Bonferonni correction
Statistical Analysis 2: Comparison: Placebo vs 20 cc of 0.5% Ropivacaine; Test type: Superiority or Other; p = 0.003, Dunns test; Median Difference (Net) = 10, 95% CI 2-sided [3 to 15]
Statistical Analysis 3: Comparison: Placebo vs 20 cc of 0.25% Ropivacaine; Test type: Superiority or Other; p = 0.14, Dunns test; Mean Difference (Net) = 5, 95% CI 2-sided [-1 to 12]

ADVERSE EVENTS:
Arm/Group | Placebo | Study Drug | 20 cc of 0.25% Ropivacaine
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Ropivacaine blood levels were not obtained. Distribution of study drug unable to gauge due to general anesthesia. Study underpowered to detect a difference in opioid consumption or global QoR-40 between the ropivacaine 0.25% and 0.5% groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No